CLINICAL TRIAL: NCT06943079
Title: Effects of Hold-relax Technique With or Without Blood Flow Restriction on Pain, Range of Motion and Functional Disability in Patients With Post Operative ACL Rehabilitation.
Brief Title: PNF and BFR Affect on Pain, ROM & Functional Outcome in Post-op ACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0120
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Sports Physical Therapy
Keywords: ACL reconstruction; Hamstring graft; Hold relax technique; Blood flow restriction; Knee joint

STUDY DESIGN:
Intervention Model Description: 2 groups; A for the application of HRT B includes HRT and BFR Their effects will be noted on 0 week, 3rd week and 6th week to conclude its result.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Hold Relax technique with Blood Flow Restriction technique (Experimental): Effects of Hold Relax technique with Blood Flow Restriction on functional outcome
  Interventions: Device: Effect of Hold Relax technique with Blood Flow Restriction technique on functional outcome
- B - Hold relax technique without blood Flow Restriction technique (Active Comparator): Effect of Hold Relax technique without Blood flow restriction on functional outcomes
  Interventions: Other: Effect of Hold Relax technique without Blood Flow Restriction technique on functional outcomes

INTERVENTIONS:
Device: Effect of Hold Relax technique with Blood Flow Restriction technique on functional outcome — Participants are randomly allocated to group A through computerised generated method. The both combine intervention is divided into 3 intervals and their results will be calculated on 0 week, 3rd, and 6th week. On every interval, pain through numeric pain rating scale, range of motion through goniometer, and functional disability through lower extremity functional scale will be measured. 2-3/week frequency of intervention will be applied on the participant.
  Other Names: Hold Relax teachnique; Blood Flow Restriction technique
  Arms: A - Hold Relax technique with Blood Flow Restriction technique
Other: Effect of Hold Relax technique without Blood Flow Restriction technique on functional outcomes — Participants are randomly allocated to group B through computerised generated method. The intervention is divided into 3 intervals and their results will be calculated on 0 week, 3rd, and 6th week. On every interval, pain through numeric pain rating scale, range of motion through goniometer, and functional disability through lower extremity functional scale will be measured. 2-3/week frequency of intervention will be applied on the participant.
  Other Names: Hold Relax technique
  Arms: B - Hold relax technique without blood Flow Restriction technique

SUMMARY:
A randomized controlled trial investigated the effects of Hold Relax Technique (HRT) with and without Blood Flow Restriction (BFR) on pain, range of motion (ROM), and functional disability in patients with post-operative ACL rehabilitation. This study includes all types of genders with age limit is 25-45 years. But the aim is to infer the answers to the following questions; Does HRT has better effects than HRT with BFR? How much effect should be noted ? The research will show that if both HRT and HRT with BFR groups had significant pain reduction, the HRT with BFR group demonstrated greater ROM improvement and significant enhancement in functional ability compared to the HRT and control groups.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted under Riphah International University guidelines and nonprobability convenient sampling will be used to collect data from the 48 participants from the Ghurki trust and teaching hospital setting. Participants will go through ACL reconstruction specifically the usage of a hamstring graft. The participants were allocated into two groups by using randomization through computer-generated software A and B. In A group only HRT will be applied to check the effects on pain, ROM, and functional disability. In the B group HRT with BFR will be utilized to note the effects on pain, ROM, and functional disability.

ELIGIBILITY:
Inclusion Criteria:

* Age group 25-45 years.
* Both gender male and female.
* Patient underwent arthroscopic ACL repair procedure.
* Patients in 6 weeks of rehabilitation phase.
* Grafts of hamstring muscle were used in repair.
* Max range achieved after post-op day 1.
* Low- moderate pain intensity.

Exclusion Criteria:

* Any form of bone carcinoma.
* Any Post-OP active infectionous Patients.
* Any circulatory effects.
* DVT and pulmonary embolism.
* Loose Implant placement.
* Non co-operative Patient.
* Hyperasthetic Patient.
* Polytraumatic Post-OP Patient.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
1- BFR Cuff | 6 weeks
  BFR requires a tourniquet to be placed on a limb. The cuff needs to be tightened to a specific pressure that occludes venous flow while still allowing arterial flow whilst exercises are being performed. Simple pieces of equipment such as surgical tubing or elastic straps have been used in gym settings to achieve this result. These are not advisable as you are unable to monitor the amount of blood flow occlusion. A thin diameter may also cause too much local pressure and result in tissue damage.(29)
2- UNIVERSAL GONIOMETER | 6 weeks
  The measurement of joint range of motion (ROM), also referred to as goniometry, is a crucial physical therapy practice.(30) Goniometry, the measuring of joint angles, is a frequently used assessment tool in the tracking of rehabilitation interventions as well as issues with the musculoskeletal system. It is generally performed with a universal goniometer (UG).(31) Inter-tester reliability for universal goniometers is mediocre.(32)
3- NUMERIC PAIN RATING SCALE (NPRS) | 6 weeks
  The Numeric Pain Rating Scale (NRS-11) is an eleven-point rating system with a score of 0 representing no pain at all and a score of 10 representing the greatest agony the patient has ever had. In this context, the NPRS-11 pain severity score of "4" is usually given particular weight, indicating that it may serve as a threshold value for pain severity in clinical practice.(33) Its dependability coefficient is high (0.95-0.96).(34)

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar Senior Lecturer, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Ghurki Trust and Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Chesworth BM, Culham E, Tata GE, Peat M. Validation of outcome measures in patients with patellofemoral syndrome. J Orthop Sports Phys Ther. 1989;10(8):302-8. doi: 10.2519/jospt.1989.10.8.302. PMID 18796951
- [Background] Kujala UM, Jaakkola LH, Koskinen SK, Taimela S, Hurme M, Nelimarkka O. Scoring of patellofemoral disorders. Arthroscopy. 1993;9(2):159-63. doi: 10.1016/s0749-8063(05)80366-4. PMID 8461073
- [Background] Irrgang JJ, Snyder-Mackler L, Wainner RS, Fu FH, Harner CD. Development of a patient-reported measure of function of the knee. J Bone Joint Surg Am. 1998 Aug;80(8):1132-45. doi: 10.2106/00004623-199808000-00006. PMID 9730122
- [Background] Martin DP, Engelberg R, Agel J, Swiontkowski MF. Comparison of the Musculoskeletal Function Assessment questionnaire with the Short Form-36, the Western Ontario and McMaster Universities Osteoarthritis Index, and the Sickness Impact Profile health-status measures. J Bone Joint Surg Am. 1997 Sep;79(9):1323-35. doi: 10.2106/00004623-199709000-00006. PMID 9314394
- [Background] McHorney CA, Tarlov AR. Individual-patient monitoring in clinical practice: are available health status surveys adequate? Qual Life Res. 1995 Aug;4(4):293-307. doi: 10.1007/BF01593882. PMID 7550178
- [Background] Nelson EC, Berwick DM. The measurement of health status in clinical practice. Med Care. 1989 Mar;27(3 Suppl):S77-90. doi: 10.1097/00005650-198903001-00007. PMID 2646493
- [Background] Al-Hadidi F, Bsisu I, AlRyalat SA, Al-Zu'bi B, Bsisu R, Hamdan M, Kanaan T, Yasin M, Samarah O. Association between mobile phone use and neck pain in university students: A cross-sectional study using numeric rating scale for evaluation of neck pain. PLoS One. 2019 May 20;14(5):e0217231. doi: 10.1371/journal.pone.0217231. eCollection 2019. PMID 31107910
- [Background] Bergh A, Lauridsen NG, Hesbach AL. Concurrent Validity of Equine Joint Range of Motion Measurement: A Novel Digital Goniometer versus Universal Goniometer. Animals (Basel). 2020 Dec 19;10(12):2436. doi: 10.3390/ani10122436. PMID 33352686
- [Background] Perez-de la Cruz S, de Leon OA, Mallada NP, Rodriguez AV. Validity and intra-examiner reliability of the Hawk goniometer versus the universal goniometer for the measurement of range of motion of the glenohumeral joint. Med Eng Phys. 2021 Mar;89:7-11. doi: 10.1016/j.medengphy.2021.01.005. Epub 2021 Jan 27. PMID 33608127
- [Background] Keil H, Beisemann N, Swartman B, Schnetzke M, Vetter SY, Grutzner PA, Franke J. Intraoperative revision rates due to three-dimensional imaging in orthopedic trauma surgery: results of a case series of 4721 patients. Eur J Trauma Emerg Surg. 2023 Feb;49(1):373-381. doi: 10.1007/s00068-022-02083-x. Epub 2022 Sep 1. PMID 36048181
- [Background] Dong HY, Tong MS, Wang J, Liu Y, Tao GY, Petersen RH, Jara-Palomares L, Wang Y, Sun YB, Chen J. Risk factors for pulmonary embolism in lung cancer patients with lower limb deep venous thrombosis: a case-control study. Transl Lung Cancer Res. 2023 Jul 31;12(7):1539-1548. doi: 10.21037/tlcr-23-346. Epub 2023 Jul 19. PMID 37577319
- [Background] Muller S, Buhl L, Nuesch C, Pagenstert G, Mundermann A, Egloff C. Favorable Patient-Reported, Clinical, and Functional Outcomes 2 Years After ACL Repair and InternalBrace Augmentation Compared With ACL Reconstruction and Healthy Controls. Am J Sports Med. 2023 Oct;51(12):3131-3141. doi: 10.1177/03635465231194784. Epub 2023 Sep 7. PMID 37675973
- [Background] Barman SR, Chan SW, Kao FC, Ho HY, Khan I, Pal A, Huang CC, Lin ZH. A self-powered multifunctional dressing for active infection prevention and accelerated wound healing. Sci Adv. 2023 Jan 25;9(4):eadc8758. doi: 10.1126/sciadv.adc8758. Epub 2023 Jan 25. PMID 36696504
- [Background] Rim CH, Park S, Yoon WS, Shin IS, Park HC. Radiotherapy for bone metastases of hepatocellular carcinoma: a hybrid systematic review with meta-analyses. Int J Radiat Biol. 2023;99(3):419-430. doi: 10.1080/09553002.2022.2094020. Epub 2022 Aug 8. PMID 35758976
- [Background] Ayres JM, Dallman J, Nolte JA, Higginbotham N, Baker J, Horton G, Salava J, Sojka J, Templeton KJ, Malancea RI, Heddings A. Managing Post-Operative Pain in Orthopedic Patients: An International Comparison. Kans J Med. 2023 Feb 21;16(1):56-60. doi: 10.17161/kjm.vol16.18744. eCollection 2023. PMID 36845259
- [Background] Helito CP, da Silva AGM, Sobrado MF, Guimaraes TM, Gobbi RG, Pecora JR. Small Hamstring Tendon Graft for Anterior Cruciate Ligament Reconstruction Combined With Anterolateral Ligament Reconstruction Results in the Same Failure Rate as Larger Hamstring Tendon Graft Reconstruction Alone. Arthroscopy. 2023 Jul;39(7):1671-1679. doi: 10.1016/j.arthro.2023.01.101. Epub 2023 Feb 10. PMID 36774971
- [Background] Kotsifaki R, Korakakis V, King E, Barbosa O, Maree D, Pantouveris M, Bjerregaard A, Luomajoki J, Wilhelmsen J, Whiteley R. Aspetar clinical practice guideline on rehabilitation after anterior cruciate ligament reconstruction. Br J Sports Med. 2023 May;57(9):500-514. doi: 10.1136/bjsports-2022-106158. Epub 2023 Feb 2. PMID 36731908
- [Background] Buckthorpe M, Gokeler A, Herrington L, Hughes M, Grassi A, Wadey R, Patterson S, Compagnin A, La Rosa G, Della Villa F. Optimising the Early-Stage Rehabilitation Process Post-ACL Reconstruction. Sports Med. 2024 Jan;54(1):49-72. doi: 10.1007/s40279-023-01934-w. Epub 2023 Oct 3. PMID 37787846
- [Background] Li S, Shaharudin S, Abdul Kadir MR. Effects of Blood Flow Restriction Training on Muscle Strength and Pain in Patients With Knee Injuries: A Meta-Analysis. Am J Phys Med Rehabil. 2021 Apr 1;100(4):337-344. doi: 10.1097/PHM.0000000000001567. PMID 33727516
- [Background] Korkmaz E, Donmez G, Uzuner K, Babayeva N, Torgutalp SS, Ozcakar L. Effects of Blood Flow Restriction Training on Muscle Strength and Architecture. J Strength Cond Res. 2022 May 1;36(5):1396-1403. doi: 10.1519/JSC.0000000000003612. Epub 2020 Apr 13. No abstract available. PMID 32287091
- [Background] Early KS, Rockhill M, Bryan A, Tyo B, Buuck D, McGinty J. EFFECT OF BLOOD FLOW RESTRICTION TRAINING ON MUSCULAR PERFORMANCE, PAIN AND VASCULAR FUNCTION. Int J Sports Phys Ther. 2020 Dec;15(6):892-900. doi: 10.26603/ijspt20200892. PMID 33344005
- [Background] Cayco CS, Labro AV, Gorgon EJR. Hold-relax and contract-relax stretching for hamstrings flexibility: A systematic review with meta-analysis. Phys Ther Sport. 2019 Jan;35:42-55. doi: 10.1016/j.ptsp.2018.11.001. Epub 2018 Nov 3. PMID 30423500
- [Background] Jack RA 2nd, Lambert BS, Hedt CA, Delgado D, Goble H, McCulloch PC. Blood Flow Restriction Therapy Preserves Lower Extremity Bone and Muscle Mass After ACL Reconstruction. Sports Health. 2023 May;15(3):361-371. doi: 10.1177/19417381221101006. Epub 2022 Jun 27. PMID 35762124
- [Background] Yuan J, Wu L, Xue Z, Xu G, Wu Y. Application and progress of blood flow restriction training in improving muscle mass and strength in the elderly. Front Physiol. 2023 Mar 24;14:1155314. doi: 10.3389/fphys.2023.1155314. eCollection 2023. PMID 37035674
- [Background] Jacobs E, Rolnick N, Wezenbeek E, Stroobant L, Capelleman R, Arnout N, Witvrouw E, Schuermans J. Investigating the autoregulation of applied blood flow restriction training pressures in healthy, physically active adults: an intervention study evaluating acute training responses and safety. Br J Sports Med. 2023 Jul;57(14):914-920. doi: 10.1136/bjsports-2022-106069. Epub 2023 Jan 5. PMID 36604156
- [Background] Colapietro M, Portnoff B, Miller SJ, Sebastianelli W, Vairo GL. Effects of Blood Flow Restriction Training on Clinical Outcomes for Patients With ACL Reconstruction: A Systematic Review. Sports Health. 2023 Mar-Apr;15(2):260-273. doi: 10.1177/19417381211070834. Epub 2022 Feb 8. PMID 35130790
- [Background] Labata-Lezaun N, Llurda-Almuzara L, Gonzalez-Rueda V, Lopez-de-Celis C, Cedeno-Bermudez S, Banuelos-Pago J, Perez-Bellmunt A. Effectiveness of Blood Flow Restriction Training on Muscle Strength and Physical Performance in Older Adults: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2022 Sep;103(9):1848-1857. doi: 10.1016/j.apmr.2021.12.015. Epub 2022 Jan 10. PMID 35026149
- [Background] Nishimura H, Yamaura K, Stetzelberger VM, Garcia AR, Hollenbeck JFM, Brown JR, Mologne MS, Uchida S, Philippon MJ. Biomechanical Comparison of Proximal Hamstring Reconstruction Using Distal Hamstring Graft Versus Fascia Lata Graft for Treatment of Chronic Hamstring Injury. Am J Sports Med. 2023 Dec;51(14):3756-3763. doi: 10.1177/03635465231206464. Epub 2023 Nov 17. PMID 37975438
- [Background] Minoli C, Travi M, Monti C, Ferrua P, Puce M, Radaelli S, Menon A, Tassi AL, Randelli PS. A fast, easy and reliable method for hamstrings graft size prediction in anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2023 Oct;31(10):4430-4436. doi: 10.1007/s00167-023-07510-z. Epub 2023 Jul 19. PMID 37468620
- [Background] Aagaard P, Simonsen EB, Andersen JL, Magnusson SP, Bojsen-Moller F, Dyhre-Poulsen P. Antagonist muscle coactivation during isokinetic knee extension. Scand J Med Sci Sports. 2000 Apr;10(2):58-67. doi: 10.1034/j.1600-0838.2000.010002058.x. PMID 10755275
- [Background] Gillquist J, Hagberg G, Oretorp N. Arthroscopy in acute injuries of the knee joint. Acta Orthop Scand. 1977;48(2):190-6. doi: 10.3109/17453677708985134. PMID 868504
- [Background] Konda SR, Davidovitch RI, Egol KA. Open knee joint injuries--an evidence-based approach to management. Bull Hosp Jt Dis (2013). 2014;72(1):61-9. PMID 25150328
- [Background] KAPLAN EB. Some aspects of functional anatomy of the human knee joint. Clin Orthop. 1962;23:18-29. No abstract available. PMID 14453729